CLINICAL TRIAL: NCT04196218
Title: Driving After Arthroscopic Rotator Cuff Repair or Shoulder Arthroplasty
Brief Title: Driving After Shoulder Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hawkins Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00095486
Record Dates: First submitted 2019-12-09; First posted 2019-12-12 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Shoulder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Driving assessment (Other): All subjects will undergo a driving assessment(s) following shoulder surgery.
  Interventions: Other: Driving simulator

INTERVENTIONS:
Other: Driving simulator — Computer simulated driving assessment

SUMMARY:
Patients undergoing a shoulder arthroplasty or rotator cuff repair will be enrolled in the study. Patients will be asked to undergo driving simulator assessments post-operatively in ATI Physical Therapy for up to 12 weeks after surgery in order to determine when it may be safe for them to return to driving. Additional assessments include patient-reported outcomes, range of motion, and strength measures, which are all standard of care. Study participation concludes when the patient passes the driving simulator test.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing either Rotator Cuff Repair or Shoulder arthroplasty from participating surgeon
2. Patients receiving physical therapy from ATI Patewood clinic
3. Must be able and willing to complete all study assessments and to be followed for the full course of the study.
4. Must be able to read, write and follow instructions in English.
5. In the opinion of the investigator, is that they subject is competent to participate in study activities
6. Prior to injury, patient was routinely driving.

Exclusion Criteria:

1. Prior shoulder surgery in the last 90 day
2. Individuals with a history of any underlying neurological conditions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Driving Assessment | surgery through 12 weeks post-op
  Clinical Driving Simulator

SECONDARY OUTCOMES:
Range of Motion | surgery through 12 weeks post-op
  Measuring shoulder range of motion
Strength | surgery through 12 weeks post-op
  Measuring shoulder strength
Visual Analog Pain Score | surgery through 12 weeks post-op
  Patient reported level of pain on a scale of 0 to 10, with 10 being extreme pain and 0 being no pain
Single Alpha Numeric Evaluation of the shoulder | surgery through 12 weeks post-op
  Percentage of normal for affected shoulder between 0 and 100, with 100 being a perfectly "normal" shoulder and 0 being a completely "abnormal" shoulder
Veterans Rand 12 Item Health Survey | surgery through 12 weeks post-op
  Patient reported quality of life. Score contains a physical component and mental component score. Both scales are continuous and values range from 0 to 70, with higher scoring indicating higher physical and mental component scores
Brief Resilience Scale | surgery through 12 weeks post-op
  Patient reported resilience on a scale of 0 to 30, with 30 indicating high resilience and 0 indicating low resilience
Shoulder function | surgery through 12 weeks post-op
  Shoulder function as measured by American Shoulder and Elbow Surgeons assessment